CLINICAL TRIAL: NCT01916135
Title: PET Imaging of Cancer Patients Using [18F]-SKI-249380, a Radiolabeled Dasatinib-Derivative
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-182
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Carcinoma; Sarcoma; Myeloma; Lymphoma; Melanoma
Keywords: [18F]-SKI-249380; PET Imaging; CT Imaging; 12-182
MeSH Terms: conditions — Carcinoma; Sarcoma; Neoplasms, Plasma Cell; Lymphoma; Melanoma | interventions — Blood Specimen Collection

ARMS (1):
- [18F]-SKI- 249380 and PET/CT scanning (Experimental): Patients will receive an injection of up to 7.5 (0.5-7.5) mCi of [18F]-SKI- 249380, followed by serial PET/CT scanning and blood draws, over a period of 3.5 hours, on a single day. PET scans will be performed immediately, at approximately 90 minutes, and optionally at approximately 3 hours after injection of the radiotracer. Each patient will be offered the opportunity to repeat the 18F-SKI-249380 injection and subsequent set of post-injection PET-CT scans, once, on a separate date. Each patient may or may not be receiving treatment with dasatinib therapy at the time of 18F-SKI-249380 PET, for their first PET study, as well as repeat PET study, at the discretion of their oncologist according to best clinical judgment.
  Interventions: Radiation: [18F]-SKI-249380; Procedure: PET/CT scan; Other: Blood draws

INTERVENTIONS:
Radiation: [18F]-SKI-249380
Procedure: PET/CT scan — PET scans will be performed immediately, at approximately 90 minutes, and optionally at approximately 3 hours after injection of the radiotracer. This includes an initial 30-minute PET scanning period, performed. At each subsequent time-point, a 30 minute axial body image is acquired. Images will be acquired on a state-of-the-art PET-CT scanner. A 30-45 minute scanning time-period is typical for clinical PET studies. A low-dose CT will be obtained immediately-prior to PET imaging, at each time-point.
Other: Blood draws — Blood will be drawn at the multiple time points for pharmacokinetic & metabolite analyses of 18F-SKI-249380. We anticipate these time points to be approximately 1, 5, 15, 30, and 90 minutes and 3 hours (optional), post-injection.

SUMMARY:
This study is the first time that a new experimental drug called [18F]-SKI-249380 is being used in people. [18F]-SKI-249380 is not a therapeutic drug. [18F]-SKI-249380 is a drug that will be used with PET scanners to 'see' where [18F]-SKI-249380 goes in the body, after its injected. The researchers believe that scans with [18F]-SKI-249380 might be able to find tumors in patients.

This study is being done to see how long [18F]-SKI-249380 stays in the blood, when it is given to people in tiny amounts by an injection into a vein in their arm, and to see where [18F]-SKI-249380 goes in the body. If the results of this trial are good, then the study doctors plan to use [18F]-SKI-249380 in another trial to see if scans with [18F]-SKI-249380 are better for finding tumors compared to the standard types of scans that doctors use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of histologically-confirmed neoplasm of any of the following classifications: solid malignancy, myeloid neoplasm, lymphoid neoplasm.
* Histology confirmed by MSKCC Department of Pathology.
* Disease that is either:

  * Radiologically-measurable or evaluable as defined by tumor response criteria from an MSKCC-IRB approved clinic research protocol.
  * Detectable by biopsy (eg, bone marrow) and/or peripheral blood assays obtained within 6 weeks of study enrollment
* Age between 21-90
* Negative serum pregnancy test for females of child-bearing age (11-55 years) and potential (ie, women who were not postmenopausal before the start of ongoing treatment, if applicable; and who have not had a surgical intervention whose intent or effect is sterilization, such as tubal ligation or hysterectomy.)
* Not breast-feeding, if applicable.

Exclusion Criteria:

* Refusal or inability to discontinue medications or other substances (eg, foods or dietary supplements) that may affect [18F]-SKI-249380 metabolism. Notably, as dasatinib metabolism is CYP3A4-dependent, the metabolism of [18F]-SKI-249380 may be altered by inhibitors and inducers of cytochrome P450 isoenzyme CYP3A4. The acceptability of medications and other substances used by the patient will be determined by the study investigators.
* Inability or refusal to have at least one peripheral intravenous line for intravenous access (as applicable to the day of [18F]-SKI-249380 injection and blood draws.)
* Refusal or inability to tolerate the scanning procedure (e.g., due to claustrophobia)
* Hepatic: from assays obtained <2 weeks prior to study enrollment
* Bilirubin > 1.5 x institutional upper limit of normal (ULN)
* AST/ALT >2.5 x ULN
* Albumin < 2 g/dl
* GGT > 2.5 x ULN IF Alkaline phosphatase > 2.5 x ULN.
* Renal: Creatinine >1.5 x ULN or creatinine clearance < 60 mL/min, from assays obtained <2 weeks prior to study enrollment
* Acute major illness (e.g., unstable cardiovascular condition, etc.)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | approximately 1, 5, 15, 30, and 90 minutes and 3 hours, post-injection
  This will be evaluated by non-invasive blood- and PET-based assays, at multiple time points. Blood/plasma assayed by standard radio-HPLC and/or TCA methods for quantitating activity, metabolites, and plasma protein binding will be performed.

SECONDARY OUTCOMES:
metabolism | approximately 1, 5, 15, 30, and 90 minutes and 3 hours, post-injection
  This will be evaluated by non-invasive blood- and PET-based assays, at multiple time points. Blood/plasma assayed by standard radio-HPLC and/or TCA methods for quantitating activity, metabolites, and plasma protein binding will be performed.
biodistribution | approximately 1, 5, 15, 30, and 90 minutes and 3 hours, post-injection
  This will be evaluated by non-invasive blood- and PET-based assays, at multiple time points. Blood/plasma assayed by standard radio-HPLC and/or TCA methods for quantitating activity, metabolites, and plasma protein binding will be performed.
radiation dosimetry | approximately 1, 5, 15, 30, and 90 minutes and 3 hours, post-injection
  This will be evaluated by non-invasive blood- and PET-based assays, at multiple time points. Blood/plasma assayed by standard radio-HPLC and/or TCA methods for quantitating activity, metabolites, and plasma protein binding will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dunphy, D.O., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/